CLINICAL TRIAL: NCT07321054
Title: Comparative Effects of Cervical Stabilization and Isometric Neck Exercises on Pain, Disability, Quality of Life and Kinesiophobia in Eyeglass Wearers With Non-specific Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: Comparative Effects of Cervical Stabilization and Isometric Neck Exercises in Eyeglass Wearers With Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibadat International University, Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIUI/RERC/ADT/2025/04/180
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain; Exercise Therapy; Isometric Exercise; Eyeglasses; Pain Measurement; Disability Evaluation
Keywords: Neck Pain; Kinesiophobia; Cervical Stabilization Exercises; Isometric Neck Exercises
MeSH Terms: conditions — Neck Pain; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This randomized controlled trial was double-blinded. Participants were randomly assigned to either the Cervical Stabilization Exercise group or the Isometric Neck Exercise group using a simple randomization (coin toss) method.
  Participants were informed that both interventions were effective physiotherapy treatments for chronic neck pain but were not told which group they belonged to. The outcome assessor, who had over fifteen years of experience, remained blinded to group allocation throughout data collection at baseline, week 2, and week 4.
  To maintain blinding, participants were instructed not to disclose their exercise details during assessment, and all data were recorded using coded identifiers (Group A or B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Neck Exercises (Active Comparator): Participants received isometric neck exercises (Isometric neck flexion, Isometric neck extension, Isometric lateral flexion and rotation), holding each movement for 10 s, and repeating each 5 times with a 5-s rest between each of them
  Interventions: Other: Isometric Neck Exercises
- Cervical Stabilization Exercises (Experimental): Participants received each neck stabilization exercises (Tucking in of chin, extending the neck, shrugging of shoulder, rolling of shoulder, retraction of scapular) in sitting position with a frequency of 15 repetitions 1 set with relaxation maintaining 6 seconds of contraction followed by 2 seconds of relaxation per repetition.
  Interventions: Other: Cervical Stabilization Exercises

INTERVENTIONS:
Other: Cervical Stabilization Exercises — Intervention Group B (Cervical Stabilization Exercises Group) Group B participants received each neck stabilization exercises (Tucking in of chin, extending the neck, shrugging of shoulder, rolling of shoulder, retraction of scapular) in sitting position with a frequency of 15 repetitions 1 set with relaxation maintaining 6 seconds of contraction followed by 2 seconds of relaxation per repetition.
  Arms: Cervical Stabilization Exercises
Other: Isometric Neck Exercises — Intervention Group A (Isometric Neck Exercises Group) Group A participants received isometric neck exercises (Isometric neck flexion, Isometric neck extension, Isometric lateral flexion and rotation), holding each movement for 10 s, and repeating each 5 times with a 5-s rest between each of them.
  Arms: Isometric Neck Exercises

SUMMARY:
The goal of this randomized controlled trial is to compare the effects of cervical stabilization exercises and isometric neck exercises on pain, disability, quality of life, and kinesiophobia in eyeglasses wearers with Non-specific chronic neck pain. Participants were randomly assigned to either Group A (Isometric Neck Exercises) or Group B (Cervical Stabilization Exercises) using a toss-and-trial method.

The intervention was provided over four weeks, with three sessions per week (total of 12 sessions):

Group A (Isometric Neck Exercises): Participants performed isometric neck flexion, extension, lateral flexion, and rotation. Each movement was hold for 10 seconds, repeated 5 times, with a 5-second rest between repetitions.

Group B (Cervical Stabilization Exercises): Participants performed chin tucks, neck extensions, shoulder shrugging, shoulder rolling, and scapular retractions in a sitting position. Each exercise was performed 15 repetitions, 1 set, holding a 6-second contraction followed by 2 seconds of relaxation per repetition.

DETAILED DESCRIPTION:
Non-specific neck pain, a common disorder of the musculoskeletal system, frequently manifests as discomfort and stiffness in the lateral and posterior aspects of the neck, often lacking distinctive diagnostic indicators.(1) Young adults are disproportionately affected by neck pain, with a significant proportion, between 42% and 67%, experiencing episodes within a one-year period. Notably, the Global Burden of Disease Study identifies neck pain, in tandem with low back pain, as the second most prevalent cause of disability among young adults aged 20-24, resulting in substantial years lived with disability.(2) Kinesiophobia refers to an excessive and debilitating fear of physical movement, stemming from a perceived vulnerability to pain or re-injury. This phenomenon is closely linked to pain catastrophizing, a cognitive and emotional response characterized by exaggerated negative thoughts and feelings about pain. In individuals experiencing chronic pain, pain catastrophizing can lead to a vicious cycle of increased pain perception, disability, and worsening impairment. Initially, these coping mechanisms may provide temporary relief during acute pain episodes. However, when pain persists, they can become maladaptive, perpetuating a cycle of fear, avoidance, and distress.(3) Wearing eyeglasses can significantly influence head and neck posture, as the body compensates for a reduced visual field by adjusting alignment. This compensatory mechanism may lead to chronic postural changes, including forward head posture and deep neck flexor weakness. The likelihood of developing forward head posture increases with the duration of eyeglasses use, highlighting the importance of assessing visual devices as part of patient care, especially when addressing neck pain and functional limitations.

Exercise plays a vital role in managing neck pain by restoring tissue function and maintaining daily activities. Research has demonstrated that targeted exercises, such as isometric and cervical stabilization exercises, can effectively reduce pain, improve muscle performance, and enhance endurance. Neck stabilization exercises improve joint mobility, sensorimotor function, and relaxation, while isometric exercises strengthen weak muscles through proprioceptive engagement. This study aims to compare the therapeutic effects of cervical stabilization versus isometric neck exercises on pain, disability, quality of life, and kinesiophobia in eyeglass wearers with non-specific chronic neck pain, providing insights into the most effective exercise approach for this population.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 25-50 years, using any form of eyeglasses for more than 2 years, with active non-specific chronic (more than three months) neck pain with pain intensity ≥ 5/10 on the numeric pain rating scale were included.

Exclusion Criteria:

* Participants with cognitive impairments or limitations that could impact their ability to provide informed consent or adhere to the study protocol.
* Individuals with a history of cardiovascular, pulmonary, or endocrine disease that could pose a risk to their health during exercise.
* Participants with health conditions that may prevent them from engaging in physical activity, such as severe musculoskeletal disorders or neurological impairments.
* Individuals with red flag symptoms indicative of underlying serious pathology, such as recent trauma, infection, or malignancy.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Neck Pain | Assessment was done at baseline, Week 2 and Week4
  Pain was measured by NPRS
Disability | Assessment was done at baseline, Week 2 and Week4
  Disability was measured by Neck Disability Index
Kinesiophobia | Assessment was done at baseline, Week 2 and Week4
  Kinesiophobia was measured by Tempa Scale-11

SECONDARY OUTCOMES:
Quality of life of Patients having Neck pain | Assessment was done at baseline, Week 2 and Week4
  Quality of life was measured by SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Nazim Farooq, PhD-PT, Principal Investigator — Ibadat International University
Locations (1):
- Faculty of Allied Health & Biological Sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asiri F, Reddy RS, Tedla JS, ALMohiza MA, Alshahrani MS, Govindappa SC, Sangadala DR. Kinesiophobia and its correlations with pain, proprioception, and functional performance among individuals with chronic neck pain. PLoS One. 2021 Jul 8;16(7):e0254262. doi: 10.1371/journal.pone.0254262. eCollection 2021. PMID 34237105
- [Background] Jahre H, Grotle M, Smedbraten K, Dunn KM, Oiestad BE. Risk factors for non-specific neck pain in young adults. A systematic review. BMC Musculoskelet Disord. 2020 Jun 9;21(1):366. doi: 10.1186/s12891-020-03379-y. PMID 32517732
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399